CLINICAL TRIAL: NCT02236130
Title: Peripheral Nerve Blocks in Pediatric Orthopedic Patients: Are There Any Post Recovery Benefits?
Brief Title: Peripheral Nerve Blocks in Pediatric Orthopedic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor response rate on follow up of patients
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Madhankumar Sathyamoorthy, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2014-0027
Record Dates: First submitted 2014-08-25; First posted 2014-09-10 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Pediatric Extremity Fracture; Pediatric Extremity Soft Tissue Injury
Keywords: pediatric regional
MeSH Terms: interventions — Anesthesia, General; Hydrocodone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General (Active Comparator): General Anesthesia only
  Interventions: Procedure: General Anesthesia; Drug: Opioids Morphine; Drug: Oral pain medication Acetaminophen with Hydrocodone
- Regional (Experimental): General Anesthesia combined with regional block
  Interventions: Procedure: Regional block; Procedure: General Anesthesia; Drug: Local Anesthetic Ropivacaine; Drug: Opioids Morphine; Drug: Oral pain medication Acetaminophen with Hydrocodone

INTERVENTIONS:
Procedure: Regional block — Single shot peripheral nerve block
  Arms: Regional
Procedure: General Anesthesia — General Anesthesia with O2/N2O/Sevoflurane
Drug: Local Anesthetic Ropivacaine — 0.5% Ropivacaine
  Arms: Regional
Drug: Opioids Morphine — Morphine
Drug: Oral pain medication Acetaminophen with Hydrocodone — Acetaminophen with Hydrocodone

SUMMARY:
Context:

Single shot peripheral nerve blocks have limited duration of action depending on the local anesthetic agent used in the block. But it rarely lasts longer than 12 hrs. Patients need oral analgesics at home once the block wears off to control the pain.

Objectives:

Primary Objective

To determine if peripheral nerve blocks have any advantage in terms of decreasing oral analgesic requirements in the post operative period even after the effects of the block have worn off

Secondary Objective

To determine if inclusion of single shot regional technique improves patient/family satisfaction with post operative pain management .

Study Design:

Prospective randomized single blinded study.

Inclusion Criteria

* Children aged between 6 yr and 17yr scheduled for ambulatory peripheral orthopedic surgery with moderate to severe postoperative pain.
* Surgery of moderate duration (<2hr)
* Surgery associated with minimal blood loss or fluid shifts (<10% total blood volume)
* American Society of Anesthesiologists (ASA) classification 1 or 2
* Parents able to understand follow up instructions and are able to reach at home by phone

Exclusion Criteria

* Known allergy to local anesthetics
* Preexisting neuropathy with sensory or motor deficits
* Skin infection at site of needle placement
* Parents refusal for peripheral nerve blocks

DETAILED DESCRIPTION:
80 children between the ages of 6yr and 17 yrs. scheduled for ambulatory peripheral orthopedic procedures in the operating rooms of Batson Children's Hospital will be enrolled in the study. Written informed consent will be obtained from the parents or legal guardian and assent will be obtained from patients when possible.

Once enrolled in the study, patients will be randomly assigned to one of two groups General anesthesia only (GA group) and General Anesthesia combined with regional anesthesia (RA group). Once the patients are brought to the operating room standard ASA monitors will be applied. After mask induction with O2/Nitrous oxide(N2O)/Sevoflurane(Sevo), a peripheral intravenous line will be inserted and secured. Additional IV medication propofol 2-3mg/kg will be given prior to insertion of appropriate size laryngeal mask airway (LMA). Patients in GA group will undergo the procedure under general anesthesia with Sevo/O2. Patients in the RA group will receive a peripheral nerve block appropriate for the procedure after induction of general anesthesia with O2/N2O/Sevo. The attending anesthesiologists will perform the nerve block under ultrasound guidance (Sonosite machine with high frequency probe) using 22G stimulating needle under aseptic precautions. 0.5% ropivacaine up to a total dose of 3mg/kg will be used for the block.

Anesthesia is maintained in both groups with O2/Sevo titrated to minimum alveolar concentration (MAC of) 1.5 . After surgical incision, doses of 0.05mg/kg morphine is given IV every 5 min as needed titrated to HR and BP within 10% change from baseline.

Additional IV morphine at the dose of 0.05mg/kg will be given every 10 minutes in the recovery room (PACU) as needed for pain ( Visual Analog score -VAS score >4). Total morphine consumption, length of recovery room stay and side effects such as nausea or vomiting will be recorded in the PACU.

The patients in the study will be given the following

1. A prescription for oral analgesics (lortab: hydrocodone 5mg with acetaminophen 325mg).
2. A handout about the nerve block and post op care (for patients in RA group)
3. A handout depicting the visual analog scale
4. Data sheet with date, time, pain scale and pain meds , satisfaction scale, documentation of side effects along with a stamped return envelope.

The parents will be educated about assessing pain and visual analog scale score. The parents will be instructed to give one or two pills depending on the weight (one pill for weight <50kg and 2 pills for weight >50kg)every 4-6 hrs. as needed for pain (VAS score more than 2).

The patients will be followed by phone by research nurse blinded to the group on postoperative day 2 and day 8. They will be asked about the total use of analgesics at the end of day 2 (first 48hrs) and day 7. Family satisfaction on a scale of 1 to10, Incidence of other side effects such as nausea, vomiting, sleep disturbance, feeding difficulty and prolonged numbness or motor block will also be collected.

The parents will also be requested to return the data sheet in the stamped return envelope to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 yr and 17yr scheduled for ambulatory peripheral orthopedic surgery with moderate to severe postoperative pain.
* Surgery of moderate duration (<2hr)
* Surgery associated with minimal blood loss or fluid shifts (<10% total blood volume)
* ASA classification 1 or 2
* Parents able to understand follow up instructions and are able to reach at home by phone

Exclusion Criteria:

* Known allergy to local anesthetics
* Preexisting neuropathy with sensory or motor deficits
* Skin infection at site of needle placement
* Parents refusal for peripheral nerve blocks

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: madhankumar sathyamoorthy, MBBS, MS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Segerdahl M, Warren-Stomberg M, Rawal N, Brattwall M, Jakobsson J. Children in day surgery: clinical practice and routines. The results from a nation-wide survey. Acta Anaesthesiol Scand. 2008 Jul;52(6):821-8. doi: 10.1111/j.1399-6576.2008.01669.x. Epub 2008 May 21. PMID 18498436
- [Background] Dorkham MC, Chalkiadis GA, von Ungern Sternberg BS, Davidson AJ. Effective postoperative pain management in children after ambulatory surgery, with a focus on tonsillectomy: barriers and possible solutions. Paediatr Anaesth. 2014 Mar;24(3):239-48. doi: 10.1111/pan.12327. Epub 2013 Dec 11. PMID 24330523
- [Background] Brasher C, Gafsous B, Dugue S, Thiollier A, Kinderf J, Nivoche Y, Grace R, Dahmani S. Postoperative pain management in children and infants: an update. Paediatr Drugs. 2014 Apr;16(2):129-40. doi: 10.1007/s40272-013-0062-0. PMID 24407716
- [Background] Bosenberg A. Benefits of regional anesthesia in children. Paediatr Anaesth. 2012 Jan;22(1):10-8. doi: 10.1111/j.1460-9592.2011.03691.x. Epub 2011 Sep 7. No abstract available. PMID 21895855
- [Background] Polaner DM, Martin LD; PRAN Investigators. Quality assurance and improvement: the Pediatric Regional Anesthesia Network. Paediatr Anaesth. 2012 Jan;22(1):115-9. doi: 10.1111/j.1460-9592.2011.03708.x. Epub 2011 Sep 27. PMID 21951324
- [Background] Ecoffey C, Lacroix F, Giaufre E, Orliaguet G, Courreges P; Association des Anesthesistes Reanimateurs Pediatriques d'Expression Francaise (ADARPEF). Epidemiology and morbidity of regional anesthesia in children: a follow-up one-year prospective survey of the French-Language Society of Paediatric Anaesthesiologists (ADARPEF). Paediatr Anaesth. 2010 Dec;20(12):1061-9. doi: 10.1111/j.1460-9592.2010.03448.x. PMID 21199114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General | Regional
Started | 22 | 27
Completed | 15 | 15
Not Completed | 7 | 12
Not completed — Lost to Follow-up | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General | Regional | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 27 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.55 [6 to 15] | 11.41 [6 to 15] | 11.02 [6 to 15]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Hydrocodone Dose (mg/kg)
Time Frame: day 2 and day 8 after the surgery
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | General | Regional
Number analyzed (Participants) | 15 | 15
mg/kg
  Day 2 Total hydrocodone use in mg/kg | 1.22 (0.67) | 1.36 (0.49)
  Day 8 Total hydrocodone use in mg/kg | 1.45 (0.82) | 2.15 (1.38)

2. Secondary Outcome: Patient/Family Satisfaction With Pain Management
Description: Patient/family satisfaction on a scale of 1 to 10 with 1 least satisfied and 10 completely satisfied. Family will complete the form and return to the primary investigator at the end of day 8 after surgery in the prepaid envelope provided to them at the time of the surgery.
Time Frame: one week after the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | General | Regional
Number analyzed (Participants) | 11 | 12
Participants | 10 | 11

ADVERSE EVENTS:
Arm/Group | General | Regional
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/27
Other Adverse Events (participants affected / at risk) | 0/22 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No